CLINICAL TRIAL: NCT04200898
Title: Clinical Investigation of the Cheetah System For The Correction of Myopic Refractive Errors With and Without Astigmatism
Brief Title: Clinical Investigation of the Cheetah System For The Correction of Myopia With and Without Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHTA-104-ILEX
Record Dates: First submitted 2019-12-04; First posted 2019-12-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Cheetah System: Phase 1 (Experimental): For each subject, surgeons will create an iLEX refractive correction using the investigational Cheetah femtosecond laser (either Beta 2a or Cheetah Production Equivalent [ELITA] models) and Cheetah patient interface (regular or small diameter designs) on one eye and the fellow eye may undergo a commercial refractive correction at the discretion of the investigator.
  Interventions: Device: Cheetah System
- Cheetah System: Phase 2 (Experimental): For each subject, surgeons will create an iLEX refractive correction using the investigational Cheetah femtosecond laser (either Beta 2a or ELITA models) and Cheetah patient interface (regular or small diameter designs) on one/both eyes (worse eye first followed by second eye, approximately 1 week later) based on refractive correction needs.
  Interventions: Device: Cheetah System
- Cheetah System: Phase 3 (Experimental): For each subject, surgeons will create an iLEX refractive correction using the investigational Cheetah femtosecond laser (either Beta 2a or ELITA models) and Cheetah patient interface (regular or small diameter designs) on one/both eyes (on the same day) based on refractive correction needs.
  Interventions: Device: Cheetah System

INTERVENTIONS:
Device: Cheetah System — For each subject, surgeons will create an iLEX refractive correction using the investigational Cheetah femtosecond laser (Models Cheetah Beta 2a, Cheetah Production Equivalent [ELITA]) and Cheetah patient interface (regular or small diameter designs).

SUMMARY:
This study will be a 3-phase, 12-months, prospective,single arm, multicenter, open-label, non-comparative, clinical investigation conducted at up to 7 sites. Up to 20 subjects will be enrolled in phase I, up to 30 subjects in phase II, and up to 200 subjects in phase 3 to achieve up to 350 treated eyes.

DETAILED DESCRIPTION:
Phase I will be used to evaluate performance (safety, ease of lenticule removal, procedure workflow, and software settings). During phase I (limited to partially sighted eyes as defined in the inclusion section), one eye of each subject will undergo iLEX treatment and the fellow eye may undergo a commercial refractive correction at the discretion of the investigator, provided there is at least 1.00 D of sphere refractive error based on manifest refraction. During phase I, treatment will be up to -11.00 D sphere with no astigmatism correction.

Phase II will be used to evaluate initial safety and effectiveness. During phase II, no astigmatism correction will be performed unless cyclotorsion correction after docking is available. For the first 10 subjects in phase II, iLEX treatment will be performed on one eye (worse eye) and approximately 1 week later, if treatment is warranted, on the fellow eye. Prior to second eye treatment in the first 10 subjects, subjects will be asked if they have any eye disturbances and whether they are willing to have their second eye treated in the study. Following eligible second eye treatment of the first 10 consecutive phase II subjects with no operative concerns by the investigator and medical monitor, subsequent phase II subjects may undergo iLEX treatment in both eyes on the same day.

Phase III will be used to evaluate long term safety and effectiveness (i.e., 12 months). During phase III, subjects may undergo iLEX treatment in both eyes on the same day.

ELIGIBILITY:
Inclusion Criteria:

Note: All criteria apply to each Cheetah treated eye

* Age ≥18 years old at the time of consenting.
* Subjects with refractive error within the following ranges:

  * Phase I: Partially sighted eyes (as defined below)
  * Phase II: Refractive error range in the Cheetah-treated eye/s between -2.00 D to -6.00 D and astigmatism up to -1.00 D based on manifest refraction at optical infinity. If cyclotorsion correction after docking is available, astigmatism greater than -1. 00 D can be included, provided that spherical equivalent (SE) is up to -6.00 D.
  * Phase III: Myopic refractive error in the study eye up to -12.00 D spherical equivalent (SE) and astigmatism up to - 6.00 D based on manifest refraction at optical infinity.
* Anticipated residual corneal stromal thickness of at least 250 microns based on preoperative corneal pachymetry minus maximum lenticule thickness to be extracted.
* Uncorrected visual acuity of 20/40 or worse in Phase II and III subjects.
* Distance Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better for phase II and III subjects. For phase I subjects, BSCVA and pin-hole acuity of the iLEX treated eye is worse than 20/50, with at least a 2-line difference between the iLEX treated eye and the fellow eye.

Note: Potential phase I subjects to be evaluated on a case-by-case basis for interocular difference in visual acuity and enrollment to be confirmed through Medical Monitor and PI consensus.

* BSCVA ≥2 lines better than distance Uncorrected Visual Acuity (UCVA). Not applicable for phase I subjects.
* Less than or equal to 0.75 D difference between cycloplegic and manifest refraction sphere. Not applicable for phase I subjects.
* A stable refractive error (based on a previous exam, medical records, lensometry, or prescription at least 12 months prior to the preoperative manifest refraction), as defined by a change of ≤1.00 D in MRSE. Additionally, the astigmatic axis must also be within 15 degrees for eyes with >0.50 D of preoperative and historical manifest cylinder.
* Any subject eye with a history of contact lens wear within the last 4 weeks must demonstrate refractive stability according to the following:

  * Rigid contact lenses (toric or spherical) must be removed for at least 4 weeks and soft contact lenses (toric or spherical) for at least 2 weeks prior to the first refraction used to establish stability.
  * Two consecutive manifest refractions and keratometry readings must be conducted at least 7 days apart.
  * Refractive stability is defined as a change of not more than 0.50 D in manifest refractive sphere and cylinder as well as keratometry meridian (either axis) between measurements. If the subject/eye meets the refractive stability criteria, contact lens wear is not permitted prior to surgery, as specified above for rigid and soft contact lens wearers.
* Willing and capable of complying with follow-up examinations for the duration of the study.
* Signed informed consent or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment.

Exclusion Criteria:

Note: All criteria apply to each eye

* Concurrent use of systemic (including inhaled) medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment. NOTE: The use of inhaled or systemic corticosteroids, whether chronic or acute, is deemed to adversely affect healing and subjects using such medications are specifically excluded from eligibility. History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders), lupus, and rheumatoid arthritis.
* Subjects with history of Diabetes Mellitus of 12 years or more and HbA1c measurement greater than 7% within a month prior to treatment.
* Subjects with a cardiac pacemaker, implanted defibrillator or other implanted electronic device.
* History of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, symptomatic blepharitis, recurrent corneal erosion, history or evidence of corneal ulcer (including but not limited to presence of visible corneal scar, abnormal topography is NOT necessary), clinically significant dry eye syndrome, neovascularization > 1 mm from limbus), retinal detachment/repair, clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm and visible on topography. Note: For phase I subjects (partially sighted eyes), history of intraocular surgery (including cataract extraction), retinal detachment/repair, and clinically significant lens opacity is acceptable for inclusion in the study.
* Evidence of glaucoma regardless of medication regimen or control, an IOP greater than 21 mmHg at screening or propensity for narrow angle glaucoma.
* NOTE: Phase I subjects with end-stage glaucoma and completely extinguished visual field are eligible to participate in the study.
* Evidence of keratoconus, pellucid marginal degeneration, corneal dystrophy or irregularity, unstable (distorted/not clear) corneal mires on central keratometry images, corneal edema, corneal lesion, hypotony, or abnormal topography. Corneal thickness less than 470 microns at the thinnest point
* Known sensitivity or inappropriate responsiveness to any of the medications used in the postoperative course.
* Either eye does not meet all inclusion criteria and does not fall within approved indications for treatment using femtosecond or excimer Laser. Not applicable for phase I subjects.
* Desire for monovision correction. Not applicable for phase I subjects.
* Women who are pregnant, breast-feeding, or intend to become pregnant during the study.
* Participation in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Monocular Uncorrected Visual Acuity | 1 month
  Phase II and Phase III effectiveness endpoint. The proportion of eyes with each acuity line of Uncorrected Visual Acuity will be summarized at 1 month postoperative visit.
maintenance of Best Spectacle Corrected Visual Acuity | 12 months
  Phase II and III primary safety endpoint.The proportion of eyes with Best Spectacle Visual Acuity acuity line changes from preoperative visit will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision
Locations (6):
- Svjetlost Eye Clinic, Zagreb, City of Zagreb, Croatia
- India (2):
  - Narayana Nethralaya Eye Hospital, RajajiNagar, Bangalore
  - Centre For Sight, New Delhi, National Capital Territory of Delhi
- Centro Oculistico Bresciano, Brescia, Italy
- Singapore (2):
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital PTE. LTD., Singapore

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu